CLINICAL TRIAL: NCT05733728
Title: Retrospective Register for Uveal Melanoma
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, Ophthalmologist, Medical University of Vienna
Other Study IDs: 1942/2022
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uveal Melanoma
  Interventions: Other: any therapy suitable

INTERVENTIONS:
Other: any therapy suitable — any therapy suitable

SUMMARY:
Background: Uveal melanoma (UM) is a common primary ocular malignancy associated with limited overall survival in the advanced stage of the disease. Fundamental breakthrough regarding the management of the disease and the overall-survival have not yet been achieved. Studies with large cohorts are difficult to perform due to limited patient numbers, therefore retrospective analyses are of great potential to gain further knowledge in a disease with high clinical needs.

Aim: The proposed project is a register for patients with UM treated at the Department of Ophthalmology and Optometry at the Medical University of Vienna between 01.01.1997 and 31.12.2021.

Patients and Methods: Patients treated for UM at the Department of Ophthalmology and Optometry at the Medical University of Vienna between 01.01.1997 and 31.12.2021 will be included in the register. Information on the baseline characteristics, survival times and course of the disease will be gathered via retrospective chart review and saved in a password-secured database.

ELIGIBILITY:
Inclusion Criteria

* Patients 18 - 99 years
* Diagnosis of uveal melanoma Exclusion Criteria
* Patients younger than 18 years of age
* Inadequate or missing information on the clinical course in patient charts

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uveal melanoma
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Conduction of a Register providing the basis for | 1997-2021
  Retrospective studies analyzing the obtained data and easy identification of patients for prospective studies (e.g. long-term survival analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No